CLINICAL TRIAL: NCT02078323
Title: Investigation of Linaclotide's Effect on the Bi-directional Brain and Gut Axis in IBS-C Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Satish Rao, Principal Investigator, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: LNZ-IT-01
Record Dates: First submitted 2014-01-08; First posted 2014-03-05 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Irritable Bowel Syndrome With Constipation (IBS-C)
Keywords: Irritable Bowel Syndrome with Constipation (IBS-C); Linaclotide
MeSH Terms: interventions — linaclotide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Linaclotide (Active Comparator): Linaclotide 290micrograms q day 30 min before meal for a 10 week period
  Interventions: Drug: Linaclotide
- placebo (Placebo Comparator): Placebo q day 30 min before meal for a 10 week period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Linaclotide
  Arms: Linaclotide
Drug: Placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to understand how a drug called Linaclotide improves bowel function and abdominal pain in patients with Irritable Bowel Syndrome with Constipation (IBS-C) as well as to examine whether Linaclotide alters communication between the brain and pelvic-floor region.

Linaclotide has been shown to improve abdominal pain and bowel symptoms in IBS-C, and is approved by the FDA for the treatment of this condition. However, how exactly this drug works to relieve abdominal pain and discomfort in humans is not clearly known. Studies in animal models suggest that patients with IBS-C have hypersensitivity in the gut.

Consequently, in IBS-C patients, there is rapid and excessive conduction of signals both from the brain and central nervous system region towards the pelvic-floor (anorectal axis) and the reverse direction. The investigators hypothesize that treatment with Linaclotide may improve/normalize these signals and thereby improve bowel symptoms.

Investigators will test this theory using a new, noninvasive (and established) method of studying this communication pathway between the brain and gut.

DETAILED DESCRIPTION:
modulate these mechanisms and thereby improve visceral pain.

Investigators propose three specific aims:

1. Examine the hyperexcitability of the afferent-pelvic floor brain axis in 60 patients with IBS by measuring the cortical evoked potentials (CEP) and sensory thresholds after electrical stimulation of the rectum and anus before and after administration of linaclotide or placebo for a period of 10 weeks.
2. Study the efferent brain pelvic floor axis by stimulating the cortex with transcranial magnetic stimulation and record the anal and rectal motor evoked potentials (MEP) in 60 IBS-C patients.
3. Determine the locus for neuronal modulation i.e are the neuroenteric changes due to central or peripheral neuronal sensitization or both, by evoking anal and rectal MEPs after selectively stimulating the lumbar and sacral nerves bilaterally, and by comparing segmental with transcranial-induced MEPs.

ELIGIBILITY:
Inclusion Criteria:

* During the previous year, all patients must have recurrent abdominal discomfort or pain for at least 3 days per month in the last 3 months associated with two or more of the following symptoms (36): i) improvement with defecation; ii) onset associated with a change in frequency of stool; and/or iii) onset associated with a change in form (appearance) of stool.
* No evidence for structural diseases- (excluded by colonoscopy, sigmoidoscopy or barium enema). Patients over 50 will not be eligible to enroll unless they have had a colonoscopy, sigmoidoscopy or barium enema within ten years prior to screening. Individuals under the age of 50 would only be required to undergo one of such diagnostic procedures if they present with alarm symptoms such as rectal bleeding, unexplained weight loss or anemia). There is no plan undergo such procedures as part of this research protocol. Therefore, individuals requiring such a procedure will be referred back to their treating physician (due to reaching age 50 and requiring a general screening of colon check or any age, due to alarm symptoms) and will not be enrolled in the study.
* No evidence of metabolic problems (to be excluded by laboratory testing; a comprehensive blood count and metabolic panel are required to be within six months of screening visit. If none are available on the patient's electronic records or records provided by an external provider, we will have them complete blood testing to exclude clinically significant metabolic abnormalities). The P.I. will decide if any values that fall out of range represent clinical significance or not.
* Women of childbearing potential must agree to a urine pregnancy test at screening and to avoid pregnancy throughout the study.
* On a prospective symptom/stool diary patients reported i) presence of abdominal pain/discomfort for at least 2 days per week; ii) hard or lumpy stools >25% and loose or watery stools in < 25% of bowel movements (IBS-C); (iii) loose or watery stools in >25% of bowel movements and hard stools <25% of Bowel Movements(IBS-D); >25% of hard or loose stools within one week (IBS-M)

Exclusion Criteria:

* Patients with laxative abuse, anorexia nervosa, and bulimia;
* Patients taking opioids (e.g. codeine or morphine), antispasmodics (dicyclomine or hyoscyamine), or muscle relaxants (e.g. cyclobenzaprine). If a patient is taking any of these drugs or supplements, and the P.I. determines that they may be able to safely come off of their medication, the patient may be eligible to re-screen, pending a two week minimum washout before enrollment;
* Patients with active episodic major depression will not be enrolled and will be referred for treatment, if necessary. Patients with a history of depression and have achieved stable remission are eligible.
* Patients with comorbid illnesses, severe cardiac disease, chronic renal failure or previous gastrointestinal surgery except cholecystectomy and appendectomy;
* Patients with neurologic diseases (e.g. head injuries, epilepsy, multiple sclerosis, strokes, spinal cord injuries) or brain disorders prone to causing seizures;
* Patients experiencing impaired cognizance (mini mental score of < 15) and/or legally blind;
* Women who are pregnant or likely to conceive (women with potential for pregnancy must use contraceptive measures to be included);
* Patients with ulcerative and Crohns colitis;
* Patients with rectal prolapse, anal fissure, anal surgery or inflamed hemorrhoids. Patients found to have any of these conditions are not eligible for enrollment due to the potential discomfort of probe placement. If a patient who is excluded due to anal fissure or inflamed hemorrhoids achieves full remission after the initial screening, they may be eligible for rescreening.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2014-02; Primary Completion 2017-10-04 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
1: Change from baseline in Prolongation and normalization of anal CEP and rectal CEP responses at 10 weeks. | at baseline assessment and at 10 weeks following baseline
  A rectal catheter will be inserted into the rectum, up to 10 cm from the anal verge. The threshold for first sensation and pain will be determined by increasing the electrical stimulation in steps of 1 mA. subsequent stimuli will be applied at an intensity of 75% of the difference between the first sensation and pain thresholds. The CEPs will be recorded in a quiet room in a semi-recumbent position. Four runs of 50 stimuli will be averaged for both the rectal and anal stimulation studies, with a 5-min rest period between each run and a 30 minute rest period between rectal and anal studies.
Change from Baseline in Prolongation and normalization of rectal MEP and anal MEP at 10 weeks. | at baseline assessment at at 10 weeks following this baseline assessment
  A 70 mm figure of eight coil, positioned over the cranium's vertex. TThe coil will be placed with the anterior edge of the cross point over the region of interest, with the handle pointing backward (for midline grid points) or at an angle of 45º tangential to the scalp surface (for lateral grid points). We will perform TMS of the anorectal motor cortex and assess the anal and rectal MEPs (EMG), by using the anorectal probe.

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University, Augusta, Georgia, United States

REFERENCES:
- [Derived] Rao SSC, Xiang X, Yan Y, Rattanakovit K, Patcharatrakul T, Parr R, Ayyala D, Sharma A. Randomised clinical trial: linaclotide vs placebo-a study of bi-directional gut and brain axis. Aliment Pharmacol Ther. 2020 Jun;51(12):1332-1341. doi: 10.1111/apt.15772. Epub 2020 May 13. PMID 32406112